CLINICAL TRIAL: NCT05896306
Title: Assessment of Cerebral Monitoring Using the Pulsatile Near Infrared Spectroscopy in Neonates Immediately After Birth - a Prospective Observational Pilot Study
Brief Title: Cerebral Monitoring Using Pulsatile Near Infrared Spectroscopy in Neonates
Acronym: pNIRS
Status: Recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 35-281 ex 22/23
Record Dates: First submitted 2023-05-31; First posted 2023-06-09 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2024-11

CONDITIONS: Neonatal Disease
Keywords: pNIRS; Neonates; Postnatal transition
MeSH Terms: conditions — Infant, Newborn, Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Term neonates
  Interventions: Other: No intervention
- Preterm neonates
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The transition from fetus to newborn is a complex physiological process. Monitoring this process to detect potential disruptions is critical but remains a challenge. Initial evaluation of neonates is usually based on visual inspection, palpation and/or auscultation, and response to stimuli. To objectify the condition of the newborn during this vulnerable transitional period, Virginia Apgar developed a clinical assessment-based scoring system called the Apgar Score, which is widely used around the world. However, there is significant inter-observer and intra-observer variability in clinical assessments using the Apgar score. To objectively assess the condition of the newborn, the latest guidelines for postnatal adaptation and resuscitation recommend the use of electrocardiography (ECG) and pulse oximetry in the delivery room in addition to clinical evaluation. These monitoring methods allow non-invasive continuous monitoring of SpO2 (Oxygen saturation) as well as heart rate (HR), but do not provide information about potentially compromised cardiovascular status, resulting in severely restricted oxygen transport to tissues.

Cerebral Oxygenation:

The brain is one of the most vulnerable organs to hypoxia during the postnatal adaptation period. The recommended routine monitoring during the neonatal transition is SpO2 and heart rate. Unfortunately, these parameters do not provide any information about cerebral blood flow or oxygen supply or brain activity. About 30% of premature babies develop cerebral hemorrhage in the first 3 days after birth. This can lead to the development of hydrocephalus, poor neurological outcome and even death. For the above reasons, there is increasing interest in additional brain monitoring. Our research group has already shown in various studies that additional cerebral monitoring using near-infrared spectroscopy (NIRS) is possible in newborns immediately after birth and may be beneficial during this vulnerable phase of life. Furthermore, this add-on monitoring could inform interventions to optimize brain oxygenation, potentially affecting survival with improved short- and long-term neurological outcomes.

Background:

The transition from fetus to newborn is a complex physiological process. Monitoring this process to detect potential disruptions is critical but remains a challenge. Initial evaluation of neonates is usually based on visual inspection, palpation and/or auscultation, and response to stimuli. To objectify the condition of the newborn during this vulnerable transitional period, Virginia Apgar developed a clinical assessment-based scoring system called the Apgar Score, which is widely used around the world. However, there is significant inter-observer and intra-observer variability in clinical assessments using the Apgar score. To objectively assess the condition of the newborn, the latest guidelines for postnatal adaptation and resuscitation recommend the use of electrocardiography (ECG) and pulse oximetry in the delivery room in addition to clinical evaluation. These monitoring methods allow non-invasive continuous monitoring of SpO2 as well as HR, but do not provide information about potentially compromised cardiovascular status, resulting in severely restricted oxygen transport to tissues.

Pulsatile mode of NIRS Recently, Hamamatsu developed new software and implemented it as a pulsatile mode in one of their near-infrared spectroscopy (NIRS) instruments, the NIRO 200 NX. In contrast to the conventional NIRS technique, which measures tissue saturation closer to venous oxygen saturation than arterial oxygen saturation, the pulsatile NIRS technique uses a higher measurement rate of 20 Hertz and can therefore measure cerebral pulse rate (cPR) and cerebral arterial oxygen saturation (SnO2) in small vessels.

Using the non-invasive pulsatile NIRS technique could be a viable new method to continuously monitor blood flow to the brain during resuscitation. This can be particularly beneficial for critically ill newborns and premature babies.

To date, no data have been published in neonates using the pulsatile NIRS technique.

ELIGIBILITY:
Inclusion Criteria:

* Term and preterm neonates observed routinely at the resuscitation desk
* Decision to conduct full life support
* Written parental informed consent

Exclusion Criteria:

* No decision to conduct full life support
* No written parental informed consent
* Congenital malformation

Ages: 0 Minutes to 15 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Term and preterm neonates after birth.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of cerebral oxygenation in cerebral pusatile vessels | 15 minutes
  cerebral oxygenation in pusatile vessels (SnO2)

CONTACTS AND LOCATIONS:
Locations (1):
- Division Neonatology, Dep. Pediatrics, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: Undecided